CLINICAL TRIAL: NCT03943199
Title: Randomized Clinical Trial: Comparison of Lysine Clonixinate, Ketorolac and Metamizole Sodium in Poisoning by Scorpion Stings
Brief Title: Comparison of Lysine Clonixinate, Ketorolac and Metamizole Sodium in Scorpion Stings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mexican Red Cross (Other)
Collaborators: Instituto Bioclon S.A. de C.V. (Industry)
Responsible Party: Principal Investigator, Josue Saul Almaraz Lira, Principal Investigator, Mexican Red Cross
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CRM-Alacran-2019
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Scorpion Stings; Pain; Analgesic
MeSH Terms: conditions — Scorpion Stings; Pain | interventions — Pain Measurement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Metamizole sodium (Active Comparator): 1 gram intravenous, will be diluted in 0.9% physiological solution of 100 ml, applied for 30 minutes
  Interventions: Diagnostic Test: Visual Analogue Scale for pain
- Ketorolac (Active Comparator): 60 milligrams intravenously, it will be added to 20 ml with 0.9% physiological solution, it will be applied for 5 minutes
  Interventions: Diagnostic Test: Visual Analogue Scale for pain
- Lysine Clonixinate (Active Comparator): 100 milligram intravenously, diluted in 5% glucose solution of 100 ml, applied for 30 minutes
  Interventions: Diagnostic Test: Visual Analogue Scale for pain
- Placebo (Placebo Comparator): 20 milliliters of 0.9% physiological solution, will be applied for 5 minutes.
  Interventions: Diagnostic Test: Visual Analogue Scale for pain

INTERVENTIONS:
Diagnostic Test: Visual Analogue Scale for pain — Will be assessed at 0´, 30´, 60´, 90 minutes and 18 hours after the application of the analgesic.

SUMMARY:
The cases of scorpion stings are matters of medical importance, where Mexico is considered as one of the main countries of such public health problem.

DETAILED DESCRIPTION:
The states with the highest incidence of cases in 2018 were Jalisco with 47370 bite reports, Guerrero with 40672 cases and Guanajuato with 40331, according to the national epidemiological surveillance system.

Due to the high affinity on ion channels, where a cystine inhibitor BmP01, it is directed to the nociceptive ion channel TRPV1 to produce pain.Pain has been reported to occur in approximately 97% of patients They are seen in the emergency room.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pain by scorpion stings
* Patients> 18 years old
* Clinical diagnosis of scorpion sting poisoning grade I, II and III.
* Chronic degenerative diseases (renal failure, hypertension, liver damage)

Exclusion Criteria:

* Patients who reject the continuation of medical treatment
* Patients who are transferred to a unit of second level of care.
* Patients with pharmacological treatment prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of antivenom as a pain treatment by the visual analogue scale of pain in poisoning by scorpion stings. | 18 hours after drugs in study
  Comparison of venom metabolism in patients valued at 18 hours with Visual Analog Scales (VAS) valued from 0 to 10

SECONDARY OUTCOMES:
Evaluate the analgesic efficacy of clonixinate of lysine, ketorolac and sodium metamizol, by the visual analogue scale of pain in poisoning by scorpion stings. | 0, 30, 60 and 90 minutes after administered the drug
  Comparison of the effectiveness inter group over the pain by scorpion sting by Visual Analog Scales (VAS) valued from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Luis H Chávez Haro, Study Director — Investigator; Josue Saul H Almaraz, Principal Investigator — Investigator
Locations (1):
- Cruz Roja Mexicana, Delegación León, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No